CLINICAL TRIAL: NCT03135522
Title: Pilot of Zinc Acetate to Improve Chronic Cough
Acronym: ZICO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00132534; 1R34HL132369-01 (NIH)
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Cough
Keywords: Chronic cough; Refractory cough; Chronic refractory cough; Zinc; Zinc acetate
MeSH Terms: conditions — Cough; Chronic Cough | interventions — Zinc Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zinc Acetate 50 mg oral capsule (Active Comparator): 50 mg zinc acetate oral capsules, over-encapsulated, administered starting at 1 capsule/day and escalated to 3 capsules/day by Day 8 post-randomization (if tolerated)
  Interventions: Drug: Zinc Acetate 50 Mg Oral Capsule
- Placebo oral capsule (Placebo Comparator): Placebo matched to zinc acetate 50 mg oral capsule active arm, administered starting at 1 capsule/day and escalated to 3 capsules/day by Day 8 post-randomization (if tolerated)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Zinc Acetate 50 Mg Oral Capsule — * Day 0 (randomization) to day 3 Zinc acetate 50 mg per day (one capsule)
  * Day 4 to day 7 If well tolerated: Zinc acetate 100 mg per day (two capsules)
  * Day 8 to V5 (6 weeks) If well tolerated: Zinc acetate 150 mg per day (three capsules)
  Other Names: Galzin
  Arms: Zinc Acetate 50 mg oral capsule
Drug: Placebo oral capsule — * Day 0 (randomization) to day 3 Placebo (one capsule per day)
  * Day 4 to day 7 If well tolerated: placebo (two capsules per day)
  * Day 8 to V5 (6 weeks) If well tolerated: placebo (three capsules per day)
  Arms: Placebo oral capsule

SUMMARY:
The Pilot of Zinc Acetate to Improve Chronic Cough (ZICO) is a study of 36 patients with chronic refractory cough that will be used to (1) assess if zinc acetate (150 mg/day) will improve patient reported measures of cough, (2) to establish if treatment with zinc acetate is well tolerated, and (3) to determine if the trial logistics are feasible.

DETAILED DESCRIPTION:
Chronic refractory cough in adults is defined as a cough lasting more than 8 weeks that does not resolve with treatment for asthma/eosinophilic airway disease, gastroesophageal reflux disease (GERD), or rhinosinusitis/post-nasal drip; and is not caused by smoking, angiotensin-converting-enzyme (ACE) inhibitors, or parenchymal lung disease. This is one of the most common conditions leading to specialty referral accounting for about 20% of new pulmonary consultations. Chronic refractory cough leads to severe impairment of quality of life and social isolation as well as sleep deprivation and chronic fatigue. The few available treatments have limited benefit and substantial side effects or abuse potential. While there are validated tools to measure the health-impact of chronic cough which can provide feasible clinical trial outcome measures, there have been no academic multi-center trials of chronic cough, and guidelines for treatment continue to rely largely on opinion rather than evidence. ZICO is a small scale randomized proof-of-concept clinical trial to establish the safety and tolerability of zinc in this population. The primary outcome measure will be the Cough Specific Quality of Life Questionnaire (CQLQ). Participants will be 18 years or older, with chronic cough lasting at least 3 months, which has been unresponsive to treatments for asthma, GERD or other upper airway disease. Individuals that are current smokers, use an ACE inhibitor, currently take zinc supplements (or multivitamins with zinc), or whose medical history includes primary parenchymal lung disease, congestive heart failure, chronic kidney disease, or another medical condition that could interfere with the study or are pregnant or breast-feeding will be excluded. Participants will be randomized to receive 6 weeks of treatment with either zinc acetate or placebo. Follow-up assessments will occur at 1, 3, 6 and 8 weeks after randomization; the final assessment is after a two week washout to establish the duration of treatment effect. In addition to completing a daily cough diary, participants will complete cough specific and general quality of life measures, complete spirometry testing and have serum zinc and copper levels measured.

ELIGIBILITY:
Inclusion Criteria:

* No upper or lower respiratory infection within 4 weeks
* Either

  * Negative evaluation for:

    * Asthma; no symptoms of disease or no evidence of asthma based on spirometry and/or methacholine challenge test
    * GERD: no symptoms of acid reflux disease or negative potential of hydrogen (pH) probe
    * Rhinosinusitis/upper airway cough

Or

* Cough persists despite treatment for the following:

  * Asthma -treated for at least 8 weeks with at least medium dose inhaled corticosteroids or with oral corticosteroids
  * GERD - treated for at least 8 weeks with either a proton pump inhibitor (PPI) or H2 blocker
  * Upper airway disease, postnasal drip or sinusitis - treated for at least 8 weeks with nasal steroids, antihistamines or both.

    * Non-smoker; defined as
* no smoking of any substance (e.g., tobacco, e-cigarette, marijuana) in the past 6 months, and
* less than 20 pack-year smoking history

  * Chest x-ray or CT scan in the past 12 months; negative for parenchymal lung diseases (such as interstitial lung disease, idiopathic pulmonary fibrosis, pneumonia, or TB) and negative for lung cancer
  * Overall Cough Visual Analog Scale (Cough-VAS) score of 30 or higher
  * Willing to halt use of zinc supplements or multivitamins containing zinc for the duration of the study
  * Provide written informed consent

Exclusion Criteria:

* Marijuana use (smoking or ingestion of marijuana) in the past 6 months
* Use of ACE inhibitor currently or within the past 6 weeks
* Use of zinc supplements or multivitamins containing zinc currently or within the past 6 weeks
* Occupational exposure to dust or chemicals that may cause cough, as determined by study physician
* Diagnosis or evidence of chronic obstructive pulmonary disease (COPD) as defined by forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) < 0.70 and FEV1% predicted < 80%
* History of lung disease, such as:

  * Bronchiectasis
  * Interstitial lung disease
  * Sarcoidosis
  * Pneumoconiosis
  * Asbestosis
  * Chronic mycobacterial infection
  * Lung cancer
* History of pancreatitis
* Congestive heart failure
* Chronic kidney disease (creatinine clearance < 30ml/min)
* Pregnant or breast-feeding
* Other medical conditions that would interfere with participation in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wise, MD, Principal Investigator — Johns Hopkins University; Janet Holbrook, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health
Locations (5):
- United States (5):
  - National Jewish Medical and Research Center, Denver, Colorado
  - St. Vincent Health, Indianapolis, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Zinc Acetate 50 mg Oral Capsule: 50 mg zinc acetate oral capsules, over-encapsulated, administered starting at 1 capsule/day and escalated to 3 capsules/day by Day 8 post-randomization (if tolerated)
  Zinc Acetate 50 Mg Oral Capsule: • Day 0 (randomization) to day 3 Zinc acetate 50 mg per day (one capsule)
  * Day 4 to day 7 If well tolerated: Zinc acetate 100 mg per day (two capsules)
  * Day 8 to V5 (6 weeks) If well tolerated: Zinc acetate 150 mg per day (three capsules)
- Placebo Oral Capsule: Placebo matched to zinc acetate 50 mg oral capsule active arm, administered starting at 1 capsule/day and escalated to 3 capsules/day by Day 8 post-randomization (if tolerated)
  Placebo oral capsule: • Day 0 (randomization) to day 3 Placebo (one capsule per day)
  * Day 4 to day 7 If well tolerated: placebo (two capsules per day)
  * Day 8 to V5 (6 weeks) If well tolerated: placebo (three capsules per day)
Period: Overall Study
Arm/Group | Zinc Acetate 50 mg Oral Capsule | Placebo Oral Capsule
Started | 17 | 17
Completed | 16 | 17
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zinc Acetate 50 mg Oral Capsule | Placebo Oral Capsule | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 62 [56 to 70] | 62 [48 to 67] | 62 [52 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 14 | 14 | 28
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 17 | 34
Smoking Status [Count of Participants; unit: Participants]
  Former | 2 | 3 | 5
  Never | 15 | 14 | 29
E-cigarette usage [Count of Participants; unit: Participants] | 0 | 0 | 0
Household Income, yearly [Count of Participants; unit: Participants]
  Less than $30,000 | 4 | 3 | 7
  $30,001 - 50,000 | 0 | 0 | 0
  $50,001 - 75,000 | 3 | 2 | 5
  Over $75,000 | 6 | 12 | 18
  Declined to answer | 4 | 0 | 4
Highest level of education completed [Count of Participants; unit: Participants]
  More than eighth grade but not high school grad | 0 | 1 | 1
  High school graduate or equivalent | 3 | 1 | 4
  Some college | 2 | 3 | 5
  Graduate of two year college or technical school | 3 | 0 | 3
  Graduate of four-year college | 3 | 8 | 11
  Post-graduate studies | 6 | 4 | 10
Health insurance [Count of Participants; unit: Participants]
  Private insurance | 11 | 14 | 25
  Public insurance | 5 | 3 | 8
  Don't know | 1 | 0 | 1
Cough characteristics [Count of Participants; unit: Participants]
  Cough upon awakening | 11 | 12 | 23
  Cough during the rest of the day or night | 17 | 16 | 33
  Persistent phlegm in chest | 7 | 5 | 12
Frequency of cough [Count of Participants; unit: Participants]
  Almost every day | 14 | 16 | 30
  Several days a week | 3 | 1 | 4
Has asthma based on spirometry or methacholine challenge [Count of Participants; unit: Participants] | 8 | 6 | 14
Has gastroesophageal reflux disease based on diagnosis or a positive pH probe [Count of Participants; unit: Participants] | 10 | 10 | 20
Has rhinosinusitis, postnasal drip, and/or upper airway disease [Count of Participants; unit: Participants] | 14 | 6 | 20
Cough medications [Count of Participants; unit: Participants] — Use of indicated medications for cough within the past two weeks.
  Participants
    Cough suppressants | 4 | 3 | 7
    Benzonatate | 1 | 0 | 1
    Other cough medications | 0 | 3 | 3
    None of the above | 12 | 11 | 23
Breathing medications [Count of Participants; unit: Participants] — Use of indicated medications for breathing within the past two weeks.
  Participants
    Bronchodilators | 7 | 6 | 13
    Inhaled corticosteroids | 1 | 1 | 2
    Other medications for breathing | 1 | 0 | 1
    None of the above | 8 | 10 | 18
Acid reflux medications [Count of Participants; unit: Participants] — Use of indicated medications for acid reflux within the past two weeks.
  Participants
    Proton pump inhibitors | 5 | 7 | 12
    Histamine 2 receptor blockers | 1 | 0 | 1
    Other acid reflux medications | 0 | 0 | 0
    None of the above | 11 | 10 | 21
Rhinosinusitis medications [Count of Participants; unit: Participants] — Use of indicated medications for rhinosinusitis within the past two weeks.
  Participants
    Nasal steroids | 8 | 5 | 13
    Oral antihistamines | 2 | 0 | 2
    Other runny nose or postnasal drip medications | 3 | 1 | 4
    None of the above | 4 | 11 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Cough Quality of Life Questionnaire (CQLQ) Score by Treatment Group
Description: Unadjusted comparison of change in CQLQ score between zinc acetate and placebo treatment groups. CQLQ scores range from 28 to 112, with lower scores indicating fewer adverse events. A minimum clinically importance difference of 5 has been proposed for this questionnaire.
Time Frame: Baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Zinc Acetate 50 mg Oral Capsule | Placebo Oral Capsule
Number analyzed (Participants) | 17 | 17
score on a scale | -5.00 [-14.00 to 0.00] | -6.00 [-18.00 to 0.00]

2. Secondary Outcome: Change in Leicester Cough Questionnaire (LCQ) Score by Treatment Group
Description: Unadjusted comparison of change in LCQ scores between zinc acetate and placebo treatment groups. LCQ scores range from 3 to 21, with lower scores indicating a greater impact of cough upon one's life. The minimum clinically importance difference for the LCQ for people with chronic cough is 1.3.
Time Frame: Baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Zinc Acetate 50 mg Oral Capsule | Placebo Oral Capsule
Number analyzed (Participants) | 17 | 17
score on a scale | 2.55 [1.16 to 4.13] | 2.59 [0.52 to 5.04]

3. Secondary Outcome: Change in Cough Visual Assessment Scale (C-VAS) Scores by Treatment Group
Description: Unadjusted comparison of change in overall severity of cough as measured by C-VAS between zinc acetate and placebo treatment groups. C-VAS scores cover four domains - severity of cough in daytime, nighttime, and overall, and severity of urge to cough. Scores range from 0 to 100 for each domain with overall scores ranging from 0 to 400. Lower scores indicate less severity. Overall severity of cough is the only domain reported here.
Time Frame: Baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Zinc Acetate 50 mg Oral Capsule | Placebo Oral Capsule
Number analyzed (Participants) | 17 | 17
score on a scale | -15.24 [-32.00 to -0.99] | -17.82 [-29.52 to -7.62]

4. Secondary Outcome: Change in Global Assessment of Change in Cough (GACC) Score by Treatment Group
Description: Unadjusted comparison of change in GACC scores between zinc acetate and placebo treatment groups. GACC scores measure change in quality of life related to cough in four domains - activity limitation, symptoms, emotions, and overall quality of life. GACC scores range from -3 (very much worse) to 3 (very much better).
Time Frame: Baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Zinc Acetate 50 mg Oral Capsule | Placebo Oral Capsule
Number analyzed (Participants) | 17 | 17
score on a scale | 0.50 [0.00 to 1.25] | 0.25 [0.00 to 0.75]

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Zinc Acetate 50 mg Oral Capsule | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/17 | 1/17
Other Adverse Events (participants affected / at risk) | 1/17 | 3/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zinc Acetate 50 mg Oral Capsule (N=17) | Placebo Oral Capsule (N=17)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant admitted to hospital with acute pancreatitis. Participant had prior history of pancreatitis; underwent pancreatic resection and splenectomy about 6 weeks after initial presentation.
Herniated disc (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Participant admitted to hospital for emergent back surgery to treat a herniated lumbar disc.
Urosepsis (Renal and urinary disorders) | 0 (0) | 1 (1) — Participant admitted to hospital with bronchitis, fever, and urinary tract infection; treated with oral and IV antibiotics and released. Participant had not started study medication at the time of event.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zinc Acetate 50 mg Oral Capsule (N=17) | Placebo Oral Capsule (N=17)
Skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Participant experienced rash and itching during titration phase of treatment. Participant stopped study drug and returned study drug to clinic.
Elevated copper level (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Serum copper level above upper limit of normal. Study physician informed participant of result.
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Participant developed skin rash on left arm. Rash treated with ointment prescribed by dermatologist; participant reported rash gone after 2 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT03135522/Prot_SAP_000.pdf